CLINICAL TRIAL: NCT02373865
Title: Randomized Double Blind Parallel Design Study Comparing Risk of Nocturnal Hypoglycemia and Critical Arrhythmia With Sitagliptin Versus Glimepiride in Patients With Type 2 Diabetes Insufficiently Controlled With Metformin Monotherapy
Brief Title: Risk of Nocturnal Hypoglycemia and Arrhythmias With Sitagliptin Versus Glimepiride in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Premature termination due to insufficient patient recruitement..
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIA-2-REDESIGN
Record Dates: First submitted 2015-01-08; First posted 2015-02-27 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes mellitus type 2; nocturnal hypoglycemia; metformin monotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Patients receiving Sitagliptin 100 mg+ Glimepiride-placebo (adapted dosage)
  Interventions: Drug: Sitagliptin; Drug: Glimepiride-Placebo
- Arm B (Active Comparator): Glimepiride (adapted dosage) + Sitagliptin 100 mg Placebo
  Interventions: Drug: Glimepiride; Drug: Sitagliptin-Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin will be given in a daily dosage of 100 mg
  Arms: Arm A
Drug: Glimepiride — Glimepiride will be given in a starting daily dosage of 1 mg which will be adapted up to 6 mg
  Arms: Arm B
Drug: Sitagliptin-Placebo — Sitagliptin-Placebo will be given additional to Glimepiride (blinded). It will be given in a daily dosage of 100 mg
  Arms: Arm B
Drug: Glimepiride-Placebo — Glimepiride-Placebo will be given additional to Sitagliptin (blinded). It will be given in a starting daily dosage of 1 mg which will be adapted up to 6 mg
  Arms: Arm A

SUMMARY:
This exploratory double blind randomized active controlled study is designed to assess the effects of a treatment with therapeutical dosage of sitagliptin versus therapeutical dosage of glimepiride as add on therapy in patients with diabetes mellitus type 2 (T2DM) patients inadequately controlled on metformin monotherapy.

DETAILED DESCRIPTION:
Type 2 Diabetes is associated with an increased cardiovascular morbidity and mortality. Among patients insufficiently controlled with metformin multimorbidity and polypharmacy is common that makes the patients frail for cardiovascular complications related to hypoglycemic events.

This exploratory double blind randomized active controlled study is designed to assess the effects of a treatment with therapeutical dosage of sitagliptin versus therapeutical dosage of glimepiride as add on therapy in patients with T2DM patients inadequately controlled on metformin monotherapy.

Examinations will be performed as a 5 day recording of subcutaneous glucose concentration (CGMS) and holder ECG (AMEDTEC) at baseline and after a 12 weeks treatment with sitagliptin or glimepiride as active comparators used in combination with metformin.

With recording of nocturnal hypoglycemia and arrhythmias it is aimed to evaluate favorable glycemic profile under treatment with sitagliptin compared to glimepiride. The primary objective is risk of serious HE for both drugs.

The glycemic profile of sitagliptin as add-on therapy to metformin seems to be favorable compared to sulfonylureass such as glimepiride. Treatment with sitagliptin as add-on to metformin therapy causes less glycemic fluctuations and may be associated with lower oxidative stress and down regulation of low grade inflammation. This hypothesis will be tested as an explorative double blind study.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* age 40-80 years
* stable dose of ≥ 1500 mg metformin or maximal tolerated dose of metformin for > 6 weeks
* HbA1c ≥ 7 % - ≤ 9.0% for age < 65 years and ≥ 7.5 % - ≤ 9.0% for age ≥ 65 years
* able and trained to perform SMBG
* the informed consent form must be signed before any study specific tests or procedures are done
* ability to understand and follow study-related instructions

Exclusion Criteria:

* Type 1 diabetes
* previous treatment with insulin, GLP1 analogues and SU in < 6 month
* HbA1c > 9 % or FPG > 15 mmol/l at randomization
* renal impairment with eGFR < 60 ml/min
* medical history of severe hypoglycemia defined as necessity of medical assistance in < 1 year
* major cardiovascular event (MACE) in medical history < 6 months
* preexisting atrial fibrillation, , AV block ≥II degree, pace-maker, implanted defibrillator
* major cardiovascular event in medical history < 6 months
* heart failure NYHA ≥ III
* contraindications to glimepiride and sitagliptin or to any excipients according to product information
* severe cognitive deficits
* Patients who are disable to read and understand informative aspects of the trial
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s)
* Inability to comply with study procedures
* Pregnant or breast-feeding woman and woman without adequate method of contraception

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markolf Hanefeld, Prof. Dr., Study Director — GWT-TUD GmbH
Locations (1):
- GWT-TUD GmbH / Studienzentrum Hanefeld, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the time period between the start of the clinical trial (march 2015 (approval of German competent authority) and the premature termination (Jan 2017) only 4 patients of originally planned 68 patients could be recruited. Recruitment period started at 09.11.2015 when first patient was enrolled into study.
Pre-assignment Details: no pre-assignment details are available for this study
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Sitagliptin 100 mg+ Glimepiride-placebo (Adapted Dose): Patients receiving Sitagliptin 100 mg+ Glimepiride-placebo (adapted dosage)
  Sitagliptin: Sitagliptin will be given in a daily dosage of 100 mg
  Glimepiride-Placebo: Glimepiride-Placebo will be given additional to Sitagliptin (blinded). It will be given in a starting daily dosage of 1 mg which will be adapted up to 6 mg
- Arm B: Glimepiride (Adapted Dose) + Sitagliptin 100 mg Placebo: Glimepiride (adapted dosage) + Sitagliptin 100 mg Placebo
  Glimepiride: Glimepiride will be given in a starting daily dosage of 1 mg which will be adapted up to 6 mg
  Sitagliptin-Placebo: Sitagliptin-Placebo will be given additional to Glimepiride (blinded). It will be given in a daily dosage of 100 mg
- Total: Total of all reporting groups
Arm/Group | Arm A: Sitagliptin 100 mg+ Glimepiride-placebo (Adapted Dose) | Arm B: Glimepiride (Adapted Dose) + Sitagliptin 100 mg Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (2.82) | 69 (9.89) | 64 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Germany | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Hypoglycemic Episodes (HE) Under Treatment With Sitagliptin Compared to Glimepiride
Description: measurement of hypoglycemic episodes including event duration at baseline and EOT after 12 weeks of treatment and measurement of time spent below critical values for hypoglycemic episodes are the primary objectives of this study. We will calculate overall episodes/time (5 days) and nocturnal episodes.
Time Frame: 12 weeks (at baseline and at EOT)
Population: Due to an impeded recruitment of patients the study was terminated. Between start (March 2015) and premature termination (Jan 2017) only 4 patients could be recruited. The reason for "0" Participants Analyzed provided in the Analysis Population Description is intended to report that data were not reported due to the termination of the study.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Occurence and Number of Nocturnal Ventricular Arrhythmias
Description: measurement of nocturnal ventricular arrhythmias at baseline and EOT (after 12 weeks of treatment) - per patient, couplets per patient, triplets per patient)
Time Frame: 12 weeks (at baseline and at EOT)
Population: as for outcome 1
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Glycemic Variability (Profile) of Sitagliptin Compared to Glimepiride
Description: The glycemic profile is defined as the area under the glucose-timeprofile obtained by continuous glucose monitoring (5 days baseline and 5 days after 12 weeks of each treatment)
Time Frame: 12 weeks (at baseline and at EOT)
Population: as for outcome 1
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A: Sitagliptin 100 mg+ Glimepiride-placebo (Adapted Dose) | Arm B: Glimepiride (Adapted Dose) + Sitagliptin 100 mg Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Limitations of the study: deceleration of patient recruitment, break up of patient recruitment, descriptive reporting of patient characteristics of 4 enrolled patients (no statistically reliable results are available)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes